CLINICAL TRIAL: NCT05101928
Title: Ozurdex as Monotherapy for Treatment of Non-infectious Intermediate, Posterior, or Panuveitis
Brief Title: Ozurdex Monotherapy Trial
Acronym: OM
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was withdrawn due to insufficient participant enrollment.
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Chloe Gottlieb, Primary Co-Investigator, Ottawa Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRRF ID 3008
Record Dates: First submitted 2021-10-11; First posted 2021-11-01 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Uveitis, Posterior; Uveitis, Intermediate; Panuveitis
MeSH Terms: conditions — Uveitis, Posterior; Uveitis, Intermediate; Panuveitis | interventions — Calcium Dobesilate; Vision, Ocular; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intravitreal Dexamethasone Implant Group (Experimental): Subjects randomized to the experimental group will receive a 0.7mg intravitreal dexamethasone (DEX) implant which will be injected in the vitreous cavity as one of the treatments of interest in this study.
  Interventions: Drug: Ozurdex 0.7mg Ophthalmic Implant
- Prednisone Taper Group (Active Comparator): Subjects randomized to the comparator group will receive oral prednisone. The initial dose is expected to range between 40 to 60mg of oral prednisone per day, with gradual tapering to the lowest dose that controls inflammation and eventually transitioning to a maintenance dose. Maintenance dose will be gradually lowered as per standard of care if remission is achieved for 6 to 12 months.
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Ozurdex 0.7mg Ophthalmic Implant — A 0.7mg intravitreal dexamethasone implant will be used for the treatment of posterior, intermediate and panuveitis for minimum of 6 months.
  Arms: Intravitreal Dexamethasone Implant Group
Drug: Prednisone — The comparator will be a prednisone taper which is currently the standard care for the uveitis types of focus.
  Arms: Prednisone Taper Group

SUMMARY:
This study will investigate the efficacy and safety of OZURDEX® (dexamethasone intravitreal implants; DEX, Allergan, Inc. Irvine, CA) as monotherapy for the treatment of non-infectious intermediate-, posterior- or panuveitis. This is a prospective randomized controlled clinical trial taking place at the University of Ottawa Eye Institute, Ottawa, Ontario, Canada, and other possible centers in Canada. Consecutive consenting subjects who meet inclusion/exclusion criteria will be selected to participate in this study. The subjects must have either non-infectious intermediate, posterior, or panuveitis. The subjects will be randomly chosen to be part of one of two groups; one group will receive DEX as monotherapy and the other group will receive oral prednisone. Approximately 84 eyes (42 per arm) will take part in study. The primary outcome will measure the proportion of eyes with a vitreous haze score of 0 six months post initial treatment. Secondary measures will include best corrected visual acuity (BCVA), central retinal thickness (CRT) measured by spectral-domain optical coherence tomography (SD-OCT), time to vitreous haze resolution and time to failure defined at number of months with DEX implant until an adjunct therapy is indicated. Baseline measurements will be recorded within 1 month prior to treatment in both groups, with follow up measurements collected at 0, 1, 2, 4, 6 and 12 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of non-infectious intermediate, posterior, or panuveitis in at least one eye
* Active uveitic disease at Screening/Baseline defined by the presence of at least 1 of the following parameters: 1) Active, inflammatory, chorioretinal and/or inflammatory retinal vascular lesion 2) ≥ 1+ vitreous haze (NEI/SUN criteria)

Exclusion Criteria:

* Presence of isolated anterior uveitis
* Evidence of macular edema due to diabetes, retinal vein occlusion or any other ocular conditions
* Confirmed or suspected active ocular disease or infections
* Intraocular surgery in the past 6 months
* History of glaucoma
* Intraocular pressure (IOP) of >21 mmHg at Screening/Baseline or confirmed normal-tension glaucoma
* Intravitreal or periocular injection within 6 months prior to screening.
* Unable to tolerate systemic corticosteroids
* Prior topical corticosteroid within 1 month of screening
* Prior non-steroidal anti-inflammatory, systemic steroids, or immunomodulatory therapy (e.g. methotrexate) within 1 month of screening
* For women: pregnant or breast feeding, or planning to become pregnant while enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with Vitreous Haze score of 0 at 6 months | Measurements obtained at 6 months
  This score (using NEI/SUN criteria) is used to grade intraocular inflammation based on vitreous cells and protein exudation. A lower score is indicative of less inflammation which is the goal when using either Ozurdex implant or a oral prednisone.

SECONDARY OUTCOMES:
Best Corrected Visual Acuity at various time points | Measurements obtained at: 1 month, 2 months, 4 months, 6 months, 12 months
  This score will be used to determine the functional outcome (visual acuity) with the treatments.
Proportion of patients with vitreous haze improvement by 1, and 2 units from baseline to various time points | Measurements obtained at: 1 month, 2 months, 4 months, 6 months, 12 months
  This score will be used to look at the degree of changes in the inflammation.
Time to vitreous haze score of 0 from baseline to various time points | Measurements obtained at: 1 month, 2 months, 4 months, 6 months, 12 months
  This will be used to assess if there are differences in time to achieving lowest possible inflammation amongst groups.
Anterior chamber cells/flare from baseline to various time points | Measurements obtained at: 1 month, 2 months, 4 months, 6 months, 12 months
  Using SUN grading criteria, the proportion of patients with cells grade 0, 0.5+, 1+, 2+, 3+, 4+ and flare grade of 0, 1+, 2+, 3+, 4+ will be determined at Month 6.
Change in central average thickness (µm) from baseline to various time points | Measurements obtained at: 1 month, 2 months, 4 months, 6 months, 12 months
  This score will be used to assess anatomical changes (e.g. cystoid macular edema) with treatment
Change in central average volume (in mm3) from baseline to various time points | Measurements obtained at: 1 month, 2 months, 4 months, 6 months, 12 months
  This score will be used to assess anatomical changes (e.g. cystoid macular edema) with treatment
Change in National Eye Institute Visual Function Questionnaire 25 Score | Baseline and 12mo
  This will be used to determine impact of disease on the subject's quality of life. The worst possible score is 0 while best is 100. The higher the score, the higher the subjective visual function.
Incidence of complications | Anywhere between baseline to 12 months
  Measure complication of treatment including but not limited to cataracts formation, ocular hypertension, vitreous hemorrhage, and endophthalmitis.
Percentage of patients with Vitreous Haze score of 0 at various time points | Measurements obtained at: 1 month, 2 months, 4 months, 6 months (primary outcome), 12 months
  This score (using NEI/SUN criteria) is used to grade intraocular inflammation based on vitreous cells and protein exudation. A lower score is indicative of less inflammation which is the goal when using either Ozurdex implant or a oral prednisone.

CONTACTS AND LOCATIONS:
Locations (1):
- Ottawa Hospital Research Institute - Vision Research Centre, Ottawa, Ontario, Canada